CLINICAL TRIAL: NCT00478803
Title: Conservative Aortic Valve Surgery for Aortic Insufficiency and Aneurysms of the Aortic Root
Brief Title: Conservative Aortic Valve Surgery for Aortic Insufficiency and Aneurysms of the Aortic Root. CAVIAAR
Acronym: CAVIAAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040412; 2006-A00362-49 (Other: IDRCB)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2012-07

CONDITIONS: Aortic Valve Insufficiency; Aortic Aneurysm
Keywords: Standardized surgical procedure; Aortic root aneurysm; Dystrophic aortic insufficiency; Conservative aortic valve surgery; Aortic annuloplasty; Mechanical aortic valve replacement; Sinus of Valsalva; Cardiac Surgical Procedures
MeSH Terms: conditions — Aortic Valve Insufficiency; Aortic Aneurysm; Aortic Root Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, preservation (Experimental): aortic valve surgery(Remodeling associated with a subvalvular aortic ring annuloplasty or double sub and supra valvular aortic annuloplasty)
  Interventions: Procedure: Remodeling procedure associated with a subvalvular aortic ring or double sub and supra-valvular aortic annuloplasty
- 2, Bentall (Sham Comparator): Mechanical aortic valve replacement(isolated or composite valve and graft replacement);actual surgical standard for dystrophic aortic roots
  Interventions: Device: Mechanical valve replacement (isolated or composite valve and graft replacement); actual surgical standard for dystrophic aortic roots

INTERVENTIONS:
Procedure: Remodeling procedure associated with a subvalvular aortic ring or double sub and supra-valvular aortic annuloplasty — Remodeling procedure associated with a subvalvular aortic ring: a) Five "U" stitches are placed inside out in the subvalvular plane (3 stitches 2 mm below the nadir of insertion of each cusp, 2 stitches below 2 of the 3 commissures at the base of the interleaflet triangles (no suture is placed at the base of the interleaflet triangle situated between the right and noncoronary sinuses to avoid injury of the bundle of His)); b) remodeling of the aortic root by scalloping a bulged graft (Gelweave ValsalvaTM); c) The 5 anchoring "U" stitches are passed through the inner aspect of the prosthetic aortic ring and tied down externally in the subvalvular position; d) anastomosis of the coronary ostia and to distal ascending aorta.
  Other Names: External aortic annuloplasty
  Arms: 1, preservation
Device: Mechanical valve replacement (isolated or composite valve and graft replacement); actual surgical standard for dystrophic aortic roots — Expansible Prosthetic Aortic Ring: Mechanical valve replacement (isolated or composite valve and graft replacement); actual surgical standard for dystrophic aortic roots
  Other Names: Bentall intervention
  Arms: 2, Bentall

SUMMARY:
The primary objective of the CAVIAAR study is to prove that aortic valve sparing for patients with aortic root aneurysms and/or dystrophic aortic insufficiency is associated with a 45% increase of 3 years-survival rate without increased mortality or serious increased morbidity events when compared to mechanical valve replacement.

The main hypothesis of this study is that a standardized procedure of valve sparing based on external aortic annuloplasty in patients with dystrophic aortic insufficiency and/or aortic root aneurysm increases survival rate without increased mortality or serious increased morbidity events when compared with patients undergoing mechanical aortic valve replacement.

DETAILED DESCRIPTION:
The CAVIAAR trial is a multicenter, prospective open trial. Target recruitment is 260 adults with aortic root aneurysms and/or dystrophic aortic insufficiency, enrolled in 19 french centers. Patients will undergo a standardized aortic valve sparing procedure based on aortic annuloplasty or a mechanical valve replacement (130 patients in each arm). In case of valve sparing, per-operative transoesophageal echocardiography will evaluate residual aortic insufficiency after valve repair. A conversion towards a valve replacement will be performed if residual aortic insufficiency is superior or equal to grade II.

Analysis will be on an intention-to-treat basis, completed with a per-protocol analysis. Primary endpoint will be 3-years survival free of morbidity or mortality, evaluated on a composite criterion, associating mortality; structural and non-structural valvular dysfunction, valve thrombosis, embolism, bleeding event, endocarditis, reoperations and permanent valve-related impairment. In the valve sparing group, we expect less than 5% rate of operative conversion and a significant improvement of primary endpoint. As secondary goals, quality of life and criteria of valvular coaptation will be compared between the 2 groups.

Standardization is the prerequisite for evaluation of valve sparing procedure. Aim of CAVIAAR trial is to provide evidence based medicine data for the best surgical management of patients with aortic root aneurysms and/or dystrophic aortic insufficiency.

ELIGIBILITY:
INCLUSION CRITERIA :

* Adult patients with indications for elective surgery of aortic root aneurysms (bicuspid or tricuspid valves) conformed to AHA or ESC guidelines or Adult patients with indications for elective surgery of isolated dystrophic aortic insufficiency (bicuspid or tricuspid valves) conformed to AHA or ESC guidelines
* signed informed consent

EXCLUSION CRITERIA :

* Aortic stenosis
* Acute ascending aorta dissections
* Contra-indications to oral anticoagulation in case of Arm 2 (mechanical valve)
* Life expectancy < 36 mois Contra-indication for implantation of the expansible rings in Arm 1: patients are known to have sensitivity to polyester or silicone, the aortic wall is deemed unusually thin and/or friable above the native aortic annular base or local anatomy impairs the safe implantation of the device in the subvalvular position (hypertrophic cardiomyopathy with septal obstruction of the left ventricular outflow tract, calcifications, adhesions…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2007-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
survival free of morbidity or mortality | 3 years
  Primary endpoint for the CAVIAAR trial will be 3-years survival free of morbidity or mortality, evaluated on a composite criteria, associating mortality; structural and non-structural valvular dysfunction, valve thrombosis, embolism, bleeding event, endocarditis, reoperations and permanent valve-related impairment

SECONDARY OUTCOMES:
separate analysis of each component of main endpoint composite criteria | during the 3 years
minor bleeding events | during the 3 years
Analysis of details of the operative procedures and reasons for intra-operative conversions | during the intervention and in intensive care
cardiac rhythm (sinus rhythm or not) | at per-operation andduring the intervention
quality of life (Short Form SF-36) | during the 3 years
- Cardiac imaging (echocardiographic and CT-scan or MRI): coaptation height, systolic and diastolic diameters of the aortic root at the levels of the base of the aortic annulus, sinuses of valsalva, sino-tubular junction and ascending aorta | during the surgery and if there is reintervention

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LANSAC, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital BICHAT CLAUDE BERNARD, Paris, France

REFERENCES:
- [Result] Lansac E, Di Centa I, Bonnet N, Leprince P, Rama A, Acar C, Pavie A, Gandjbakhch I. Aortic prosthetic ring annuloplasty: a useful adjunct to a standardized aortic valve-sparing procedure? Eur J Cardiothorac Surg. 2006 Apr;29(4):537-44. doi: 10.1016/j.ejcts.2005.12.055. Epub 2006 Feb 24. PMID 16500110
- [Derived] Lansac E, Bouchot O, Arnaud Crozat E, Hacini R, Doguet F, Demaria R, Leguerrier A, Jouan J, Chatel D, Lopez S, Folliguet T, Acar C, Leprince P, Langanay T, Jegaden O, Bessou JP, Albat B, Latremouille C, Fabiani JN, Fayad G, Fleury JP, Pasquet B, Debauchez M, Di Centa I, Tubach F. Standardized approach to valve repair using an expansible aortic ring versus mechanical Bentall: early outcomes of the CAVIAAR multicentric prospective cohort study. J Thorac Cardiovasc Surg. 2015 Feb;149(2 Suppl):S37-45. doi: 10.1016/j.jtcvs.2014.07.105. Epub 2014 Aug 12. PMID 25240525